CLINICAL TRIAL: NCT03689699
Title: Randomized Phase 1b/2 Study of Nivolumab or Nivolumab Plus BMS-986253 in Combination With Intermittent Androgen Deprivation Therapy in Men With Hormone-Sensitive Prostate Cancer
Brief Title: Nivolumab and BMS-986253 for Hormone-Sensitive Prostate Cancer (MAGIC-8)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mark Stein (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Mark Stein, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR7949
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: Immunotherapy; Nivolumab; BMS-986253; Degarelix; HuMax IL-8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; HuMax-IL8

STUDY DESIGN:
Intervention Model Description: The study will include a total of approximately 30 patients per arm to achieve at least 23 evaluable patients per arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab alone (Experimental): Men with hormone-sensitive prostate cancer will receive Nivolumab alone every 4 weeks for 8 weeks (2 doses), followed by Nivolumab + Degarelix every 4 weeks for 16 weeks (4 doses).
  Interventions: Drug: Nivolumab; Drug: Degarelix
- Arm B: Nivolumab plus BMS-986253 (Experimental): Men with hormone-sensitive prostate cancer will receive Nivolumab plus BMS-986253 every 4 weeks for 8 weeks (2 doses), followed by Nivolumab + BMS-986253 + Degarelix every 4 weeks for 16 weeks (4 doses).
  Interventions: Drug: Nivolumab; Drug: Degarelix; Drug: BMS-986253

INTERVENTIONS:
Drug: Nivolumab — A dose of 480mg every 4 weeks as a 30 minute IV infusion for 6 doses has been selected for this study. 6 total doses.
  Other Names: Opdivo®
Drug: Degarelix — Standard treatment at a dose of 240mg subcutaneously (SQ) as a loading dose followed by 80mg SQ every 4 weeks for 4 doses.
  Other Names: Firmagon®
Drug: BMS-986253 — BMS-986253 (also referred to as anti-IL8 mAb or HuMax IL8) is a fully human-sequence IgG1κ monoclonal antibody (mAb) directed against human interleukin-8 (IL-8). Subjects will be treated with an intravenous (IV) flat dose of 2400mg every 2 weeks.
  Other Names: HuMax IL-8
  Arms: Arm B: Nivolumab plus BMS-986253

SUMMARY:
MAGIC-8 is a two-arm, multicenter, phase 1b/2 study to assess the efficacy of immunotherapy with either Nivolumab (anti-PD-1) or Nivolumab plus BMS-986253 combined with ADT using Degarelix (LHRH antagonist) for men with hormone-sensitive prostate cancer and a rising prostate-specific antigen (PSA). The purpose of this study is to see whether immunotherapy with either Nivolumab alone or Nivolumab plus BMS-986253 combined with Degarelix, which suppresses testosterone, is safe and can decrease the chance that the cancer will come back.

The primary objectives are to 1) determine the rate of PSA recurrence defined as a PSA >0.2ng/ml for radical prostatectomy patients or PSA >2.0ng/ml for patients who received primary radiation therapy at a time point of 10 months after start of therapy; and 2) determine the safety and tolerability of either nivolumab or nivolumab plus BMS-986253 in combination with degarelix in men with hormone-sensitive prostate cancer. The secondary objectives include determining relapse-free survival (RFS) and % change in PSA to immunotherapy alone.

DETAILED DESCRIPTION:
Prostate cancer is common and remains a major cause of death in men. Following local therapy with surgery or radiation, a significant number of men recur either with a rising PSA only (biochemical recurrence (BCR)) or clear metastatic disease on imaging. Although androgen deprivation therapy (ADT) is a frequently used and effective treatment for prostate cancer, it is associated with significant side effects including fatigue, hot flashes, decreased libido and bone loss. Therefore, new approaches to decrease the time on ADT are crucial to improving quality of life for men with prostate cancer.

Once initiated, ADT can be given either continuously or intermittently. However, even with an intermittent approach the ADT-free interval typically decreases with each cycle and most men eventually develop castration resistance. Therefore new treatment strategies are needed to improve disease control while minimizing ADT exposure for men with early prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented prostatic adenocarcinoma confirmed by a pathology report from prostate biopsy or a radical prostatectomy specimen.
* Age ≥18 years
* Previously undergone primary therapy for prostate cancer. Salvage XRT or cryotherapy following primary therapy ≥ 6 months prior to randomization is allowed.
* A rising PSA defined as the following:

  * If the subject's primary therapy was RP (radical prostatectomy) (with or without adjuvant or salvage XRT), rising PSA is defined as 2 consecutive rising values above 0.2 ng/mL, each taken ≥ 3 weeks apart, and the last value ≥ 2.0 ng/mL
  * If the subject received other primary therapies (e.g. XRT, cryosurgery, brachytherapy), rising PSA is defined per the Phoenix definition, i.e., 2 consecutive rising values above the PSA nadir plus 2.0 ng/mL.
* For the biopsy sub-groups, patients must be willing to undergo pre and on- treatment biopsies.
* PSADT ≤ 12 months. PSADT(prostate-specific antigen doubling time) will be determined from all non-zero PSA values collected preferably, however not limited to, from the 12 months prior to randomization. To calculate PSADT, there must be at least THREE PSA values, with at least 4 weeks between each measurement. The PSADT will be computed from the formula: PSADT = (loge2)/k, with k being the estimated slope of the logarithm of PSA over time. The following web site may also be used: http://www.mskcc.org/applications/nomograms/prostate/PsaDoublingTime.aspx
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1, or Karnofsky score ≥ 70% (see Appendix A)
* Testosterone ≥ 150 ng/dL ≤ 28 days of prior to registration
* Adequate bone marrow, hepatic, and renal function:

  * White Blood Cell (WBC)>3,000 cells/mm3
  * Absolute neutrophil count (ANC)>1,500 cells/mm3
  * Hemoglobin >9.0 g/dL
  * Platelet count >100,000 cells/mm3
  * Serum creatinine <1.5 × upper limit of normal (ULN)
  * Serum total bilirubin <1.5 × ULN
  * ALT (alanine aminotransferase) <3 × ULN
  * AST(aspartate aminotransferase) <3 × ULN
* Willingness to provide written informed consent and HIPAA authorization for the release of personal health information, and the ability to comply with the study requirements (note: HIPAA authorization will be included in the informed consent)
* Willingness to use barrier contraception during treatment plus 5 half-lives of nivolumab (~125 days) plus 90 days (duration of sperm turnover) for a total of 215 days post-treatment completion (azoospermic men are not exempt from contraceptive requirements)

Exclusion Criteria:

Received any experimental immunotherapy on an experimental clinical trial ≤ 1 year prior to randomization

* PSA > 50 at time of enrollment
* High volume disease defined as >5 bone metastases or lymph nodes >3cm in size.
* Histologic predominance of other types of prostate cancers such as sarcomatous, lymphoma, small cell, and neuroendocrine tumors (note: a maximum of 5 subjects with ductal prostate cancer will be allowed to enroll to each arm of study treatment across all sites).
* Received salvage XRT ≤ 6 months prior to randomization
* Received ADT ≤ 6 months prior to randomization
* Received any form of chemotherapy ≤ 90 days prior to randomization
* Received granulocyte colony-stimulating factor or GM-CSF ≤ 90 days prior to randomization
* Any major surgery requiring general anesthesia ≤ 28 days prior to randomization.
* Any other concurrent or prior treatment for prostate cancer ≤ 28 days prior to randomization.
* An active infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5 o F or 38.1 o C) within 1 week prior to randomization
* Prior systemic, ongoing immunosuppressive therapy ≤ 14 days prior to study treatment administration (except for adrenal replacement steroid doses ≤ 10mgdaily prednisone equivalent in the absence of active autoimmune disease or a short course of steroids (<5 days) up to 7 days prior to initiating study treatment).
* Prior participation in an anti-IL8 clinical study
* A candidate is scheduled or likely to be scheduled for salvage external beam XRT or surgery for prostate cancer during the study period
* Concomitant treatment with other hormonal therapy or 5α-reductase inhibitors such as Dutasteride or Finasteride (prior use of these agents is allowed if ≥3 months prior to randomization).
* History of known or suspected autoimmune disease with the following exceptions:

  * Asthma and/or allergic rhinitis (seasonal allergies)
  * Vitiligo
  * Resolved childhood atopic dermatitis
  * Psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
  * Residual hypothyroidism due to an autoimmune condition only requiring hormone replacement
  * Euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin (Ig) prior to the first dose of study treatment).
  * Type 1 diabetes mellitus
* History of malignancy within the last 2 years (except non-melanoma skin cancers and superficial bladder cancer) and for which no additional therapy is required or anticipated to be required during the study period.
* Uncontrolled major active infectious, cardiovascular, pulmonary, hematologic, or psychiatric illnesses that would make the patient a poor study candidate
* Known prior or current history of HIV and/or hepatitis B/C
* Prior organ allograft

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Stein, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Weill Cornell Medical Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Sidney Kimmel Cancer Center- Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Nivolumab Alone | Arm B: Nivolumab Plus BMS-986253
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab Alone | Arm B: Nivolumab Plus BMS-986253 | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Median (Full Range); unit: years] | 68.5 [62 to 80] | 68.0 [52 to 82] | 68.3 [52 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 27 | 25 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prostate-specific Antigen (PSA) Recurrence
Description: Defined as a PSA >0.2ng/ml for radical prostatectomy patients or PSA >2.0ng/ml for patients who received primary radiation therapy at a time point of 10 months after start of therapy.
Time Frame: Up to 10 months after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab Alone | Arm B: Nivolumab Plus BMS-986253
Number analyzed (Participants) | 30 | 29
Participants | 8 | 6

2. Primary Outcome: Incidence of Adverse Events That Are Serious in Nature and Related to the Investigational Product.
Description: All participants receiving at least one dose of the study drug will be evaluated for safety and toxicity. Adverse events will be classified and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 100 days after completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nivolumab Alone | Arm B: Nivolumab Plus BMS-986253
Number analyzed (Participants) | 30 | 29
Participants | 4 | 3

3. Secondary Outcome: Percentage Change in PSA
Description: Determine the % change in PSA in response to immunotherapy by comparing the PSA prior to and following 8 weeks of immunotherapy and before initiation of ADT
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Relapse-free Survival (RFS)
Description: Relapse defined as a PSA >0.2ng/ml for radical prostatectomy patients or PSA >2.0ng/ml for patients who received primary radiation therapy.
Time Frame: Up to two years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 100 days after completion of therapy
Arm/Group | Arm A: Nivolumab Alone | Arm B: Nivolumab Plus BMS-986253
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/30 | 3/29
Other Adverse Events (participants affected / at risk) | 29/30 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab Alone (N=30) | Arm B: Nivolumab Plus BMS-986253 (N=29)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Adrenal insufficiency (Renal and urinary disorders) | 1 | 2
Autoimmune diabetes (Immune system disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pancreatitis (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab Alone (N=30) | Arm B: Nivolumab Plus BMS-986253 (N=29)
Hot flashes (General disorders) | 14 | 18
Fatigue (General disorders) | 16 | 14
Injection site reaction (Injury, poisoning and procedural complications) | 4 | 10
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 | 6
Headache (General disorders) | 1 | 4
Flu-like symptoms (General disorders) | 2 | 4
Memory impairment (General disorders) | 0 | 3
Insomnia (General disorders) | 1 | 2
Anorexia (General disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Dizziness (General disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 11
Diarrhea (Gastrointestinal disorders) | 6 | 4
Thyroid disorder (Endocrine disorders) | 7 | 5
Hepatotoxicity (Hepatobiliary disorders) | 2 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Adrenal insufficiency (Renal and urinary disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pancreatitis (Hepatobiliary disorders) | 1 | 4
Oral mucositis (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03689699/Prot_SAP_000.pdf